CLINICAL TRIAL: NCT00034814
Title: Efficacy and Safety of Talampanel as Adjunctive Therapy in Patients With Partial Seizures: A Phase II Clinical Trial.
Brief Title: Multicenter Trial for Adults With Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, Vice President, North American IR&D and Head of Global Clinical Operations, Teva Branded Pharmaceutical Products R&D, Inc.
Purpose: Treatment
Other Study IDs: IXL-201-14-189
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — talampanel

ARMS (6):
- 1 (Placebo Comparator): Enzyme-inducing placebo TID
  Interventions: Drug: Placebo
- 2 (Experimental): Enzyme-inducing Talampanel 35 mg TID
  Interventions: Drug: Talampanel
- 3 (Experimental): Enzyme-inducing TLP 50mg TID
  Interventions: Drug: Talampanel
- 4 (Placebo Comparator): Non-enzyme-inducing placebo TID
  Interventions: Drug: Placebo
- 5 (Experimental): Non-enzyme-inducing TLP 25mg TID
  Interventions: Drug: Talampanel
- 6 (Experimental): Non-enzyme-inducing TLP 35mg TID
  Interventions: Drug: Talampanel

INTERVENTIONS:
Drug: Talampanel — Non-enzyme-inducing TLP 35mg TID
  Arms: 6
Drug: Placebo — Enzyme-inducing placebo TID
  Arms: 1
Drug: Talampanel — Enzyme-inducing Talampanel 35 mg TID
  Arms: 2
Drug: Talampanel — Enzyme-inducing TLP 50mg TID
  Arms: 3
Drug: Placebo — Non-enzyme-inducing placebo TID
  Arms: 4
Drug: Talampanel — Non-enzyme-inducing TLP 25mg TID
  Arms: 5

SUMMARY:
To compare seizure frequency in patients with refactory partial seizures (with or without generalization) who are taking Talampanel versus placebo as an add-on therapy to other licensed concomitant antiepileptic drugs (AEDs) and to determine the safety of Talampanel in this group of patients.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo controlled, multicenter, efficacy and safety study of talampanel (TLP) in 190 patients (18-65 years old) with refractory partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* must weigh greater than or equal to 40kg
* Patients must have diagnosis of partial seizures
* At least 3 observable partial seizures a month
* Are currently being treated with 1 and no more than 2 marketed Anti-epileptic Drugs.

Exclusion:

* Patients on Valproic acid, and Felbamate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Reduction in frequency of partial seizures | 12 weeks
  Change in frequency of recognizable seizures as measured by entries in a seizure diary

SECONDARY OUTCOMES:
The number of seizure-free days and percent responders | 12 weeks
  A responder was defined as a patient with greater than or equal to 50% reduction in seizure frequency compared to baseline